CLINICAL TRIAL: NCT06935682
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase 1 Study to Assess the Safety and Pharmacokinetics of Y-4 Tablets After Single- and Multiple-dose in Healthy Subjects
Brief Title: Safety and Pharmacokinetics of Y-4 Tablets in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongjun Wang, Chief Physician, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y-4-LC-01
Record Dates: First submitted 2025-04-02; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adult Male and Female Volunteers
Keywords: phase I trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-4 tables (Experimental): Each subject will receive a single dose and multiple doses.
  Interventions: Drug: Y-4 tables
- Y-4 placebos (Placebo Comparator): Each subject will receive a single dose and multiple doses.
  Interventions: Drug: Y-4 placebos

INTERVENTIONS:
Drug: Y-4 tables — Each subject will receive a single dose and multiple doses. During the single dose phase (Day1-Day4), the subjects will be administered with single dose of Y-4 tablets on fasting state in the morning of Day D1. During the multiple dosing phase (Day5-Day13), the subjects will be required to administer with Y-4 tablets continuously for 6 days, BID of Day5-Day9 (once in the morning and once in the evening, Q12h) and QD of Day10, for a total of 11 doses.
  Arms: Y-4 tables
Drug: Y-4 placebos — Each subject will receive a single dose and multiple doses. During the single dose phase (Day1-Day4), the subjects will be administered with single dose of Y-4 placebos on fasting state in the morning of Day D1. During the multiple dosing phase (Day5-Day13), the subjects will be required to administer with Y-4 placebos continuously for 6 days, BID of Day5-Day9 (once in the morning and once in the evening, Q12h) and QD of Day10, for a total of 11 doses.
  Arms: Y-4 placebos

SUMMARY:
Y-4 is a new fixed-dose combination drug product containing two active ingredients of pregabalin and riluzole.

The primary objective is to evaluate the safety and tolerability of Y-4 tablets in Chinese healthy adult subjects after single- and multiple-dose.

The secondary objective is to characterize the pharmacokinetics (PK) of pregabalin and riluzole in Chinese healthy adult subjects after single- and multiple-dose of Y-4 tablets.

DETAILED DESCRIPTION:
This study will be a single-center, randomized, double-blind, placebo-controlled, dose-escalation study in Chinese healthy adult subjects. A total of 36 subjects, 3 cohorts of 12 subjects each (half men and half women), will be enrolled in this study. In each dose cohort, subjects will undergo single and multiple (BID, 11 doses) administration, among them, 10 subjects (half men and half women) will receive Y-4 tablets and 2 subjects (half men and half women) will receive placebo randomly.

After providing written informed consent, subjects will undergo screening for eligibility. Screening for the study will begin 14 days prior to the dosing. Subjects will be admitted to research center in the afternoon of Day-1 prior to the dosing day and fasting for the next 10 hours overnight. In the morning of the following day (Day 1), subjects will be administered the assigned dose of Y-4 tablets or placebo orally, then subjects will be monitored for the following 72 hours. During Day 5 to Day 9, the subjects will be required to be administered twice a day (Q12 h), once in the morning and once in the evening. In the morning of Day 10, subjects will be administered to the last dose. In the morning of Day 13 (approximately 72 hours after the last administration), the safety and tolerance will be evaluated and then subjects will be discharged.

A telephone follow-up/completion visit will be conducted 7 days (±1) post discharge.

Treatment cohorts are planned as following:

Cohort 1: 75 mg/18.75 mg Y-4 tablets (75 mg pregabalin and 18.75 mg riluzole) or placebo tablets (two little Y-4 tablets) Cohort 2: 112.5 mg/28.125 mg Y-4 tablets (112.5 mg pregabalin and 28.125 mg riluzole) or placebo tablets (one large Y-4 tablet) Cohort 3: 150 mg/37.5 mg Y-4 tablets (150 mg pregabalin and 37.5 mg riluzole) or placebo tablets (one large Y-4 tablet and one little Y-4 tablet)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female subjects, 18-45 years of age (including both ends).
2. Body weight ≥ 50 kg for male and ≥ 45 kg for female, body mass index (BMI) within the range of 19 - 28 kg/m2 (including both ends).
3. During the screening period, serum creatinine is within the normal range, or the standard creatinine clearance (CLcr) estimated by Cockcroft-Gault formula is ≥ 80 mL/min (for female subject, according to the calculation result × 0.85）.
4. Subjects who are able to understand and give their signed informed consent before any trial related procedures are performed.

Exclusion Criteria:

1. Subjects who are known to be allergic to pregabalin, riluzole or any excipients of Y-4 tablets (microcrystalline cellulose, Copovidone, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate and Opadry amb Ⅱ), have allergic diseases or allergic constitution;
2. Subjects who have special requirements for diet and cannot follow the unified diet;
3. Physical examinations, vital signs, 12-lead electrocardiograms (ECG), chest X-ray (front position), laboratory tests (hematology, serum chemistry, coagulation test, urinalysis, etc.) and other screening tests found abnormalities that the researchers judged to be of clinical significance;
4. Subjects who have experienced angioedema in the past (such as swelling of the face, mouth (tongue, lips, and gums), and neck (pharynx and throat));
5. History of dizziness or vertigo with clinical significance, or disease of inner ear known to cause dizziness or vertigo;
6. QTcF > 450 msec at the screening stage;
7. Diagnosed with insomnia, anxiety disorder, depression, epilepsy, or other serious mental disorders, and principal investigator determines that the subject is not suitable to participate in this trial;
8. Presence or history of hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of medicines;
9. Subjects who drink too much tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup = 250 mL) every day within 3 months prior to screening, or disagree that any caffeine-containing beverages are prohibited during the trial;
10. Subjects who have consume any diet (food or beverage) rich in grapefruit, pitaya, mango and cranberry within 14 days prior to screening;
11. Subjects have disease history or current disease that may affect the safety evaluation of the subject or the internal process of the study drug, including the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, immunology, psychiatry, metabolic abnormalities, gastrointestinal surgery (excluding appendicitis surgery), etc. In particular, there is a history of dysphagia or any gastrointestinal disease affecting drug absorption (including frequent nausea or vomiting caused by any cause) and eye diseases;
12. Donation or loss of blood equal to or in excess of 400 mL, or blood transfusion within 3 months prior to screening; or donation or loss of blood equal to or in excess of 200 mL within 1 month prior to screening;
13. Subjects who have taken any drugs known to be strong inhibitors or inducers of cytochrome P450 enzymes within 2 months prior to screening (such as inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors - serotonin reuptake inhibitors (SSRI) antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines); or subjects who have taken any prescription drugs, over-the-counter drugs and Chinese herbal medicine other than the above drugs within 14 days prior to screening;
14. Subjects who have taken central nervous system (CNS) depressants including opioids (pethidine hydrochloride, morphine, dihydromorphine hydrochloride, fentanyl, tramadol, etc), benzodiazepines (diazepam, flurazepam, clonazepam, oxazepam, chlordiazepine and triazolam etc), antiepileptic drugs (carbamazepine, sodium valproate, phenobarbital drugs etc) within 2 months prior to screening;
15. Subject with sleep apnea, or subjects with severe sleep snoring and daytime drowsiness;
16. Subjects with suicidal thoughts and behavior;
17. Subject participated in any other clinical trials within 3 months prior to screening;
18. Current or former drug users, or positive urine screen for drugs of abuse at screening (screening items include: dimethylenedioxyamphetamine, methamphetamine, ketamine, morphine, tetrahydrocannabinoid acid, cocaine);
19. Alcoholics or regular drinkers within 3 months prior to screening, that is, those who drink more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of alcohol with 40% alcohol content or 150 mL of wine), or whose alcohol breath test results are greater than 0.0 mg/100 mL, or who cannot abstain from alcohol during the trial;
20. Smokers or those who cannot comply with the prohibition of smoking during the trial, or positive for cotinine screening;
21. Subjects who is positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, syphilis antibody or human immunodeficiency virus (HIV) antibody;
22. Male subjects (or their partners) or female subjects have baby plans during the whole trial period and within 3 months after the end of the trial, or subjects are unwilling to take one or more non-drug contraceptive measures (such as complete abstinence, condoms, ligation, etc.) during the trial period;
23. Female subjects who have unprotected intercourse within 14 days prior to screening, or pregnant or lactating women;
24. Subjects with poor compliance or other factors unsuitable for participation in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-04 (Actual); Primary Completion 2025-05-04 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
adverse events | From the first day to the 19th± 1st day after the start of administration
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment. The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of "mild", "moderate" and "severe". The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.
Incidence of subject getting abnormal results of laboratory tests after treatment | From the first day to the 19th± 1st day after the start of administration
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Incidence of subject getting abnormal results of 12-lead ECG after treatment | From the first day to the 19th± 1st day after the start of administration
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Incidence of subject getting abnormal results of vital signs after treatment. | From the first day to the 19th± 1st day after the start of administration
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(body temperature, respiration, blood pressure, and pulse) will be assessed by according equipment.(electronic sphygmomanometer, thermometer).
Incidence of subject getting abnormal results of physical examinations after treatment. | From the first day to the 19th± 1st day after the start of administration
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation.
Incidence of subject getting abnormal results of blood oxygen saturation after treatment | From the first day to the 19th± 1st day after the start of administration
  Record changes of blood oxygen saturation from baseline to post-treatment, listing deviations from normal ranges post-treatment. Normal range is provided by the site
Incidence of subject getting abnormal results of C-SSSRS scale evaluation after treatment after treatment | From the first day to the 19th± 1st day after the start of administration
  Record changes of C-SSSRS scale evaluation from baseline to post-treatment

SECONDARY OUTCOMES:
Cmax | From day 1 to day 4 after the start of administration
  peak plasma concentration after single dose
AUC0-t | From day 1 to day 4 after the start of administration
  Area under the plasma concentration versus time curve from time 0 to the time of the last quantifiable concentration after single dose
AUC0-∞ | From day 1 to day 4 after the start of administration
  Area under the plasma concentration-time curve from time 0 to infinity (extrapolated) after single dose
Tmax | From day 1 to day 4 after the start of administration
  Time to reach maximum observed plasma concentration after single dose
t1/2 | From day 1 to day 4 after the start of administration
  Terminal elimination half-life after single dose
λz | From day 1 to day 4 and from day 8 to day 13 after the start of administration
  Terminal-phase elimination rate constant, slope of curves terminal segment at semi-log concentration-time curve calculated by linear regression.
AUC_%Extrap | From day 1 to day 4 and from day 8 to day 13 after the start of administration
  The percentage of the AUC0-inf that has been extrapolated. AUC_%Extrap = [(AUC0-∞-AUC0-t)/AUC0-∞] × 100%
CL/F | From day 1 to day 4 after the start of administration
  Total body clearance after single dose. CL/F = Dose/AUC0-inf
Vz/F | From day 1 to day 4 after the start of administration
  apparent volume of distribution after single dose. Vz/F = Dose/AUC0-∞/λz
MRT0-t | From day 1 to day 4 after the start of administration
  Mean residence time within the time from time zero to the lowest testing plasma concentration after single dose. MRT0-t = AUMC0-t/AUC0-t
MRT0-∞ | From day 1 to day 4 after the start of administration
  Mean residence time extrapolated from zero to infinity after single dose. MRT 0-∞ = AUMC 0-∞/AUC 0-∞.
Cav, ss | From day 8 to day 13 after the start of administration
  mean plasma concentration at steady state
Cmax, ss | From day 8 to day 13 after the start of administration
  Cmax at steady state
Cmin, ss | From day 8 to day 13 after the start of administration
  minimal plasma concentration at steady state
AUCτ | From 8 to day 13 after the start of administration
  Area under the concentration-time curve between dosing interval at steady state
AUC0-t, ss | From day 8 to day 13 after the start of administration
  AUC0-t at steady state
AUC0-∞, ss | From day 8 to day 13 after the start of administration
  AUC0-∞ at steady state
Tmax, ss | From day 8 to day 13 after the start of administration
  Tmax at steady state
t1/2, ss | From day 8 to day 13 after the start of administration
  t1/2 at steady state
CLss/F | From day 8 to day 13 after the start of administration
  CL/F at steady state
Vz, ss/F | From day 8 to day 13 after the start of administration
  Vz/F at steady state
DF | From day 8 to day 13 after the start of administration
  degree of fluctuation of plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No